CLINICAL TRIAL: NCT01861288
Title: Development of a New Algorithm to Determine the Activity of Disease: Deep Endoscopic Remission Assessed by a Surrogate Biomarker in Patients With IBD.
Brief Title: Deep Endoscopic Remission Assessed by a Surrogate Biomarker in Patients With Inflammatory Bowel Disease
Status: Completed | Type: Observational
Sponsor: Herlev Hospital (Other)
Collaborators: University Hospital of North Norway (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Katrine Carlsen, MD, Herlev Hospital
Other Study IDs: DER-SBIO
Record Dates: First submitted 2013-05-17; First posted 2013-05-23 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2018-02

CONDITIONS: Inflammatory Bowel Disease; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Fecal Calprotectin; Clinical IBD score (SCCAI, PUCAI, aPCDAI); Endoscopic deep remission; Histopathologic deep remission; Immunological deep remission; Treatment algorithm
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Feces
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults and children with and without IBD: The study includes adult and pediatric patients with and without IBD who, as part of an ongoing investigation or treatment, have to undergo a sigmoidoscopy (for children: colonoscopy).
  Inclusion of adult patients, age 15-67 years: 50 patients with UC in remission, 50 patients with active UC, 50 patients without IBD
  Inclusion of pediatric patients, <15 years: We expect to include: 10 UC / CD patients in remission,10 UC / CD patients in relapse,10 non-IBD patients.

SUMMARY:
We hypothesize that the number of needed endoscopic procedure performed at IBD patients (adult and children), can be reduced by using an individualized algorithm of symptoms, blood and faecal biomarkers.

The aim of the study is to reduce the numbers of endoscopies, as the procedure is uncomfortable for the patient, time consuming and expensive. Through indirect tests - blood test, fecal inflammation marker and clinical symptoms - compared to endoscopic findings, we want to construct an algorithm by which the intestinal healing can be foreseen without performing an endoscopy.

Furthermore, we will correlate FC, blood tests, clinical symptom score and endoscopic score, with the histo-pathological inflammation score from intestinal biopsies and the immunological score depicted by TNF- alpha and IL17A levels in intestinal tissue, in order to assess the gold standard - endoscopic remission.

DETAILED DESCRIPTION:
Deep remission: The treatment goal in patiens with IBD is to achieve deep remission before drug withdrawal to avoid relapse. In order to evaluate the healing of mucosa, it is currently necessary to carry out an endoscopy, despite the additional information provided by FC and blood samples. The endoscopic procedure is uncomfortable for the patient, time consuming and expensive. We therefore seek, on the basis of existing knowledge and using a correlation between FC, blood tests and clinical remission with endoscopic findings, to establish some non-invasive biomarkers that might express deep remission. In the long run, threshold levels will be used as indicators for performing an endoscopy and, hopefully, reduce the need for it to be performed. We will compare the results from children and adults because it is likely there exist differences in their respective FC levels.

Histopathologic remission: Biopsies of the intestinal tissue can be evaluated histopathologically and indicate the level of microscopic inflammation and can assess the acute and chronic inflammatory signs at the cellular level, e.g. altered glandular structure, crypt abscess and ulcerations. By using the Karl Geboes grading system, microscopic histopathological deep remission can be assessed. We will explore the endoscopic 'gold standard' by comparing endoscopic remission with histopathological remission.

Immunological remission: In general, tissue factors are linked to various immunological pathways belonging to the innate, adaptive and regulatory immune response, comprising a pro-inflammatory and an anti-inflammatory response. This includes molecules such as cytokines, chemokines, adhesion molecules and their corresponding cellular and soluble receptors. Tumor-necrosis-factor (TNF)-alpha and interleukin 17A is two of several molecules in the pro-inflammatory process that is strongly associated with the grade of inflammation in IBD (Florholmen and Fries 2011). Olsen et al. 2009 have reported that a normalization of mucosal TNF-alpha in most ulcerative colitis patients will represent an endoscopically healed mucosa.

In addition to clinical indexes, endoscopic and histological criteria, we also introduce a molecular based Immunological Remission. A working hypothesis is that immunological remission is a state of normalization of the pro-inflammatory and anti-inflammatory processes in mucosa. The concept of immunological remission and the potential clinical impact are still in the early phases of evaluation, and to obtain a practical application a non-invasive test, such as one based on a stool sample, must be developed. In the current project, immunological remission will be a part of this study, as endoscopic and histopathology remission, with correlation to FC, blood tests and clinical remission.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for endoscopy
* Age 0 - 67 years
* Intestinal infections ruled out by stool sample analysis for pathogenic bacteria, parasites and Clostridium difficile
* CMV ruled out
* Fluent in Danish

Exclusion Criteria:

* American Society of Anesthesiologists (ASA) score III or above
* Patients who are alcohol or drug abusers

Max Age: 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study includes adult and pediatric patients with and without IBD who, as part of an ongoing investigation or treatment, have to undergo a sigmoidoscopy (for children: colonoscopy).
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2013-11-01 (Actual); Primary Completion 2016-09-05 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Fecal Calprotectin (FC)and clinical score | Two FC test will be analysed up to 1 week before the endoscopy. SCCAI will be collected up to 1 week before endoscopy.
  FC is an inflammation marker from intestinal mucosa.
  Clinical score by Simple Clinical Colitis Activity Index, SCCAI. SCCAI is a specific Ulcerative Colitis index.

SECONDARY OUTCOMES:
Histopathological and Immunological inflammation score | up to 8 weeks after endoscopy
  Histopathological inflammation: intestinal biopsies assessed by Karl Geboes score.
  Immunological score: TNF- alpha and Interleukin 17 A levels in intestinal biopsies assessed by PCR analysis

OTHER OUTCOMES:
Endoscopic-, Histopathological- and Immunological- intestinal inflammation in children with IBD | Up to 2 years after endoscopy
  Comparing the results of endoscopic-, histopathological- and immunological-intestinal inflammation in children versus adults with IBD.

CONTACTS AND LOCATIONS:
Overall Officials: Katrine Carlsen, MD, Principal Investigator — Departmen of Gastroenterology, Herlev University Hospital; Pia Munkholm, Professor, Study Director — Department of Gastroenterology, Herlev University Hospital; Vibeke Wewer, MD, Phd, Study Chair — Hvidovre University Hospital; Lene Riis, MD, PhD, Study Chair — Department of Pathology, Herlev University Hospital; Christian Jakobsen, MD, PhD, Study Chair — Hvidovre University Hospital
Locations (1):
- Katrine Carlsen, Herlev, Denmark